CLINICAL TRIAL: NCT04949854
Title: Evaluating the Role of the Guidewire in Peripheral Intravenous Access: A Randomized Controlled Trial of Ultrasound-Guided Catheter Survival
Brief Title: Evaluating the Role of the Guidewire in Peripheral Intravenous Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol was substantially revised
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-049
Record Dates: First submitted 2021-06-01; First posted 2021-07-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Intravenous Vein Catheter Phlebitis; Intravenous Infection
Keywords: PIV; BBraun Ultra Long Catheter; BD Accucath; Phlebitis; IV Infection
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: This is a prospective, parallel, non-blinded, two-arm randomized (like the flip of a coin) controlled trial of catheter failure evaluating the impact of a built-in guide wire. This study plans to enroll 360 participants (two equally sized groups of 180 participants in each arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Arm B.Braun 6.35 cm 20 Gauge catheter (Active Comparator): Device 6.35 cm 20 Gauge B. Braun catheter without guidewire
  Interventions: Device: B.Braun 6.35 cm 20 Gauge ultralong intravenous catheter
- Experimental Arm B.D. Accucath 5.71 cm 20 Gauge catheter (Experimental): Device BD 5.71 cm Accucath IV catheter with guidewire
  Interventions: Device: B.D Accucath 5.71 cm 20 Gauge ultralong intravenous catheter

INTERVENTIONS:
Device: B.Braun 6.35 cm 20 Gauge ultralong intravenous catheter — control Arm 1 (6.35 cm 20 Gauge ultralong intravenous catheter without guidewire
  Arms: Control Arm B.Braun 6.35 cm 20 Gauge catheter
Device: B.D Accucath 5.71 cm 20 Gauge ultralong intravenous catheter — Experimental Arm B.D Accucath 5.71 cm 20 Gauge ultralong intravenous catheter with guide wire
  Arms: Experimental Arm B.D. Accucath 5.71 cm 20 Gauge catheter

SUMMARY:
This study is to demonstrate that the control ultralong intravenous catheter without the guide wire is equivalent to the experimental catheter with the guide wire. The hypothesis of this study is that the 6.35 cm 20G ultralong Ultrasound Guided Peripheral Intravenous (USPIV) will have no difference in survival compared to the 5.71 cm ultralong with wire USPIV.

DETAILED DESCRIPTION:
Peripheral intravenous catheter (PIVC) insertion is a standard hospital procedure that enables providers to rapidly administer fluids, medications, or blood products directly into a patients vein. This allows patients who have difficulty with tolerating oral intake or patients who are being prepared for surgery to still receive the proper treatments. Furthermore, because many medications are not designed to be administered orally, a PIVC is often used.

Despite being a common procedure, PIVC insertion routinely fails with failure rates of traditional blind intravenous (IV) catheter placement ranging from 19%-29.9%. Common causes of failure include infiltration, occlusion, dislodgement, phlebitis, and infection. In addition to increasing costs, multiple placements of an IV catheter during a hospital stay places a considerable time burden on hospital staff. One effort to alleviate this burden has been the introduction of ultrasound, which is shown to help mitigate failure rates of PIVC placement in patients with difficult vascular access. .

The catheter length in vein is the single most relevant variable in determining catheter survival in USPIV insertions. IV Catheter survival depends on the length of the catheter inside the veins. Vein depth and angle of insertion play a significant role in choosing the right catheter length to achieve the ideal quantity of catheter in vein. When a shallow angle is used, the catheter distance to the vein also increases and longer catheters are needed to achieve the optimal 2.75 cm in vein. Unfortunately, the longest most commonly stocked peripheral IV catheter at most institutions is 4.78 cm. This length is inadequate for insertions with a vein depth of greater than approximately 0.75 cm. As this is a commonly encountered vein depth, longer peripheral IV catheters are needed to ensure improved catheter survival.Few peripheral intravenous catheter options exist with the Ultra Long profile. The 6.35 cm B. Braun deep access device and the BD 5.71 cm Accucath device are two commercially available options for this category of ultra long peripheral IVs. Both catheters are available and being used in Beaumont Hospital.The 6.35 cm option is similar to other peripheral IV catheters and is inserted using the same technique applied for all ultrasound guided IV insertions. The 5.71 cm option is similar to other peripheral IVs with the additional feature of a built-in wire within the device to help guide the catheter in the vein once the needle has penetrated the vein. The cost of the 5.71 cm option is approximately ten times the cost of the 6.35 cm device.

Adult patients with a Vascular Access Score of 4 or 5 (where Score 1= Visible with distention and easily palpable; Score 2=Visible and easily palpable; Score 3= Not visible and easily palpable; Score 4=Visible and poorly palpable and Score 5=Not visible and poorly or non-palpable) will be approached for inclusion in the study.

ELIGIBILITY:
Eligible patients must be:

1. ≥ than 18 years old
2. Vascular Access Score 4 or 5.

Clinicians Eligibility Criteria:

1. Clinician working in the emergency room (physician, advanced practice provider, nurse, technician) OR clinician working on the inpatient vascular access team (advanced practice provider, nurse)
2. Greater than 6 months experience in ultrasound guided IV insertions

Patients are excluded:

1. <18 years old
2. Restricted mobility of elbow joint
3. Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Catheter survival | During hospitalization, up to 60 days
  Survival in hours or days of the catheter will be evaluated by functionality of catheter for intravenous therapy prior to patient discharge. The event of interest is failure of functionality identified during follow-up assessment during hospitalization.

SECONDARY OUTCOMES:
First-stick success. | First day of hospitalization
  Number of patients with only one puncture of skin to achieve venous access
Time to insertion | First day of hospitalization
  Time to insertion (measured in minutes) is defined as needlestick to dressing application.
Provider proficiency | Study period, a maximum of 1 year
  Change in mean number of attempts per patient for successful insertion, from baseline mean for first three patients attempted to last three patients attempted.
Total cost for all vascular access needs during hospitalization. | During hospitalization, up to 60 days
  Cost per patient for vascular access during hospitalization, comprising (i) direct costs of IV insertion based on estimated labor and material cost per insertion attempt and estimated similar costs for rescue devices if needed and (ii) cost of treatment based on estimated cost per hour.
Catheter-associated thrombosis | During hospitalization, up to 60 days
  The number of patients with all symptomatic catheter related upper extremity venous thrombosis inclusive of superficial thrombophlebitis (SVT), deep venous thrombosis(DVT), and pulmonary embolism will be confirmed by upper extremity doppler evaluation, computed tomography, and/or ventilation perfusion testing.
Catheter-associated bloodstream infection | During hospitalization, up to 60 days
  The number of patients with catheter-associated bloodstream infection. Cases of infection will be diagnosed per laboratory confirmed bloodstream infection criteria published by the National Healthcare Safety Network (NHSN) and identified by the Department of Epidemiology at Beaumont Hospital.

OTHER OUTCOMES:
Inflammatory complications by clinical assessment | During hospitalization, up to 60 days
  Number of patients with inflammatory complications measured by a score of 2 or greater on a standardized visual phlebitis scale, with a range of 0 to 5 where 0 is no inflammation and 5 is advanced stage thrombophlebitis.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD., Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospitals, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No